CLINICAL TRIAL: NCT05844475
Title: Buccal Strip Gingival Graft With a Xenogeneic Collagen Matrix Versus Free Gingival Graft for Keratinized Mucosa Augmentation at Implant Sites: A Randomized, Controlled, Clinical Trial
Brief Title: Buccal Graft + Collagen Matrix Versus Free Gingival Graft for Keratinized Mucosa Augmentation at Implant Sites
Acronym: FGGvsBSG+CM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Lorenzo Tavelli, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB23-0131
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free gingival graft (FGG) (Active Comparator): Conventional free gingival graft, involving the harvesting of an epithelialized graft from the hard palate, which is then stabilized/sutured to the recipient site (implant).
  Interventions: Procedure: Conventional Free Gingival Graft Approach (FGG)
- Buccal Strip Graft + Collagen matrix (bSG + CM) (Experimental): Strip graft obtained from the buccal mucosa of a site showing abundant keratinized gingiva, combined with a collagen matrix. The bSG + CM graft is stabilized/sutured to the recipient site (implant).
  Interventions: Procedure: Buccal Strip Graft with a collagen matrix (bSG + CM)

INTERVENTIONS:
Procedure: Conventional Free Gingival Graft Approach (FGG) — Conventional Free Gingival Graft Approach involving palatal soft tissue harvesting
  Arms: Free gingival graft (FGG)
Procedure: Buccal Strip Graft with a collagen matrix (bSG + CM) — A small strip of keratinized gingiva is harvested from the buccal gingiva of a site showing abundant keratinized gingiva, and combined with a xenogeneic collagen matrix
  Arms: Buccal Strip Graft + Collagen matrix (bSG + CM)

SUMMARY:
The study aims at comparing two different approaches for soft tissue augmentation at implants lacking keratinized and adherent mucosa width: the free gingival graft (FGG) vs the Buccal Strip Graft in combination with a xenogeneic collagen matrix (BSG + CM)

DETAILED DESCRIPTION:
Conventional free gingival graft (FGG), serving as control group, will be compared to buccal strip gingival graft (BSG) in combination with a collagen matrix (CM), serving as test group, in terms of clinical, volumetric, ultrasonographic, and patient-reported outcomes related to soft tissue augmentation at implant sites lacking keratinized and adherent mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Periodontally and systemically healthy,
* Full-mouth plaque score and full-mouth bleeding ≤ 20% (measured at four sites per tooth),
* Presence of at least one dental implant with < 2 mm of KM and lack of firm/adherent mucosa,
* Presence of at least 4 mm of keratinized gingiva in two or more teeth nonadjacent to the implant to be treated,
* Implants diagnosed as healthy (Berglundh et al. 2018),
* The patient must be able to perform good oral hygiene.

Exclusion criteria:

* Contraindications for surgery,
* Systemic condition (e.g. diabetes mellitus, HIV, cancer, etc) that could compromise wound healing,
* Patients pregnant or attempting to get pregnant (self-reported),
* Untreated periodontitis,
* Untreated peri-implant mucositis or peri-implantitis (Berglundh et al. 2018),
* Smoking,
* Allergy to collagen-based medical products or iodine,
* Previous free gingival graft procedure at the target site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Sites showing KM≥ 2 mm and AM≥ 1 mm | 6 and 12 months
  Number of sites showing at least 2 mm of keratinized mucosa width (in millimeters) and at least of 1 mm of attached mucosa (in millimeters) (outcome expressed as a number)

SECONDARY OUTCOMES:
KM width gain | 6 and 12 months
  Gain in keratinized mucosa width obtained after the intervention compared to baseline (expressed in millimeters)
AM gain | 6 and 12 months
  Gain in attached mucosa width obtained after the intervention compared to baseline (expressed in millimeters)
Mucosal thickness (MT) gain | 6 and 12 months
  Gain of mucosal thickness (MT) obtained after the intervention compared to baseline (expressed in millimeters)
Volumetric change | 6 and 12 months
  Volumetric change occurring at the treated sites analyzed by superimposing digital impressions obtained using optical scanners at baseline and 6 months (expressed in mm^3)
Ultrasonographic tissue perfusion | Baseline, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months
  Tissue perfusion changes over the healing assessed with ultrasonography (expressed in cm/s)
Post-operative morbidity | Daily, for the first 4 weeks after the procedure
  Patient-reported outcome assessed using a daily questionnaire first the first 4 weeks (expressed as a number using a 0-100 visual analogue scale [VAS])
Treatment satisfaction | 12 months
  Patient-reported outcome assessed with questionnaire including a 0-100 visual analogue scale (VAS) at the last visit (expressed as a number)
Esthetic assessment | Baseline and 12 months
  Patient-reported outcome assessed with questionnaire including a 0-100 visual analogue scale (VAS) at the initial and last visit (expressed as a number)
Ultrasonographic strain elastography | Baseline, 3 months, 6 months and 12 months
  Changes in the elasticity of the soft tissue over the healing assessed with ultrasonography (expressed as a ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Tavelli, DDS, MS, PhD, Principal Investigator — Harvard School of Dental Medicine, Boston, USA
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No